CLINICAL TRIAL: NCT03485820
Title: COMPASS: A Novel Transition Program to Reduce Disability After Stroke
Brief Title: A Novel Transition Program to Reduce Disability After Stroke
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201705047; 1R01HD092398-01 (NIH)
Record Dates: First submitted 2018-03-26; First posted 2018-04-02 (Actual); Results first posted 2025-03-05 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke; Hemorrhagic Stroke
Keywords: environmental modifications; activity performance
MeSH Terms: conditions — Ischemic Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Intervention Model Description: Single-blind, parallel-group, randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMPASS (Experimental): COMPASS is a complex intervention that combines 2 evidence-based treatment strategies at a new point of care (transition from inpatient rehabilitation). The objective of home visits by an occupational therapy (OT) practitioner is to remediate barriers in the home and community that influence daily activities and community participation. The treatment will include a set of 1 predischarge and four 75-minute postdischarge visits. The intervention is followed by 2 booster sessions.
  Interventions: Behavioral: COMPASS
- Education program (Sham Comparator): An OT practitioner will deliver the program in accordance with "Evidence-Based Educational Guidelines for Stroke Survivors after Discharge Home." Topic order is determined by participants. Four 75-minute sessions will be provided. Topics may include stroke symptoms, risk factors and preventing stroke recurrence, nutrition, managing emotions, sleep, pain. Written materials from the National Stroke Association and the American Stroke Association are provided.
  Interventions: Behavioral: Stroke education

INTERVENTIONS:
Behavioral: COMPASS — The data from the baseline assessment will be used to develop an environmental modification intervention plan. Environmental modifications will be installed before discharge if possible. Problem areas addressed are participant specific (tailored), but the process to identify and address the target area is systematic. All participants will receive identical intervention components. The standardized components include assessment, identification of problematic activities (and environmental barriers), identification of three solutions (for each problem), implementation of solution set selected by the participant, training, and active practice of daily activities in one's own home and community.
  Arms: COMPASS
Behavioral: Stroke education — The control group will experience the same effects of time and attention in the home but no effect on the outcome of interest.
  Arms: Education program

SUMMARY:
This study evaluates a program designed to help individuals transition home from inpatient rehabilitation following an ischemic or hemorrhagic stroke. Half of the participants will receive a stroke education program while the other half will receive an environmental modifications program.

DETAILED DESCRIPTION:
A gap in care exists at the point of transition from inpatient rehabilitation (IR) to home, when survivors encounter new environmental barriers due to the cognitive and sensorimotor sequelae of stroke. Resolving these barriers and improving independence in the community have potential to significantly improve stroke survivors' long-term morbidity. The proposed study investigates the efficacy and safety of a novel enhanced rehabilitation-transition program to reduce environmental barriers and improve daily activity performance and community participation.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥50 years
* acute ischemic or hemorrhagic stroke diagnosis
* independent ADLs prior to stroke (premorbid Modified Rankin Scale Score ≤2)
* plan to discharge to home

Exclusion Criteria:

* severe terminal systemic disease that limits life expectancy to < 6 months
* previous disorder (e.g. dementia) that makes interpretation of the self-rated scales difficult or Short Blessed Test (SBT) score of 10 or less (indicating significant cognitive impairment)
* moderate to severe Aphasia as determined by the NIHSS Best Language rating of 2 or more
* reside in congregate living facility.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Stark, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Krauss MJ, Somerville E, Poiter C, Bollinger RM, Holden BM, Blenden G, Kretzer D, Stark SL. Functional performance of patients with stroke during inpatient rehabilitation: a cross-sectional study of home and access visits. BMC Health Serv Res. 2025 Jan 7;25(1):34. doi: 10.1186/s12913-024-12167-6. PMID 39773227
- [Derived] Bollinger RM, Krauss MJ, Somerville EK, Holden BM, Blenden G, Hollingsworth H, Keleman AA, Carter A, McBride TD, Barker AR, Yan Y, Stark SL. Rehabilitation Transition Program to Improve Community Participation Among Stroke Survivors: A Randomized Clinical Trial. JAMA Netw Open. 2024 Oct 1;7(10):e2437758. doi: 10.1001/jamanetworkopen.2024.37758. PMID 39374016
- [Derived] Krauss MJ, Holden BM, Somerville E, Blenden G, Bollinger RM, Barker AR, McBride TD, Hollingsworth H, Yan Y, Stark SL. Community Participation Transition After Stroke (COMPASS) Randomized Controlled Trial: Effect on Adverse Health Events. Arch Phys Med Rehabil. 2024 Sep;105(9):1623-1631. doi: 10.1016/j.apmr.2024.05.015. Epub 2024 May 19. PMID 38772517
- [Derived] Somerville E, Minor B, Keglovits M, Yan Y, Stark S. Effect of a Novel Transition Program on Disability After Stroke: A Trial Protocol. JAMA Netw Open. 2019 Oct 2;2(10):e1912356. doi: 10.1001/jamanetworkopen.2019.12356. PMID 31577356

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COMPASS | Education Program
Started | 85 | 100
Completed | 77 | 66
Not Completed | 8 | 34

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COMPASS | Education Program | Total
Number analyzed (Participants) | 85 | 100 | 185
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.0) | 66.3 (9.0) | 66.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 45 | 80
  Male | 50 | 55 | 105
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 45 | 63 | 108
  White | 40 | 36 | 76
  Not listed | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 85 | 100 | 185
Marital status [Count of Participants; unit: Participants]
  Married/partner | 48 | 44 | 92
  Single/divorced/widowed | 37 | 56 | 93
Living situation [Count of Participants; unit: Participants]
  Lives alone | 26 | 32 | 58
  Lives with someone | 59 | 68 | 127
Type of stroke [Count of Participants; unit: Participants]
  Ischemic | 70 | 78 | 148
  Hemorrhagic | 15 | 22 | 37
Comorbidities [Mean (Standard Deviation); unit: number of comorbidities present] — Number of comorbidities Population: Number analyzed is lower than overall number of baseline participants due to missing data.
  number of comorbidities present
    number analyzed (Participants) | 83 | 95 | 178
    (all) | 3.5 (1.8) | 3.5 (2.3) | 3.5 (2.1)
Functional Independence Measure [Mean (Standard Deviation); unit: units on a scale] — Measurement for disability. 18 items assess six areas of function in motor ability and cognition. Final summed score ranges from 18-126: 18 represents complete dependence/total assistance, 126 represents complete independence.
  units on a scale | 76.1 (18.2) | 79.5 (18.0) | 77.9 (18.1)
Length of stay in inpatient rehabilitation [Mean (Standard Deviation); unit: days] — Population: Number analyzed is lower than overall number of baseline participants due to missing data.
  days
    number analyzed (Participants) | 85 | 98 | 183
    (all) | 20.7 (16.5) | 18.0 (7.8) | 19.3 (12.6)
Geriatric Depression Scale - Short Form score [Mean (Standard Deviation); unit: units on a scale] — 15 items assess depression among older adults. Sum score ranges from 0-15; Score >5 points is suggestive of depression. Higher scores indicate higher likelihood of depression. Population: Number analyzed is lower than overall number of baseline participants due to missing data.
  units on a scale
    number analyzed (Participants) | 84 | 96 | 180
    (all) | 3.5 (2.7) | 3.1 (2.8) | 3.3 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: Reintegration to Normal Living Index (RNLI)
Description: The RNLI is a disability-related quality-of life-instrument used to measure participants' satisfaction with their home and community participation and has been validated on a population of community-dwelling individuals with chronic conditions. It uses an 11-item, 10 point scale, with higher scores indicating greater reintegration to normal living. The sum score is divided by 110 and then multiplied by 100 to obtain an adjusted score. Adjusted scores range from 0 to 100, with higher scores indicating greater reintegration to normal living.
Time Frame: Baseline and 12 months post-stroke
Population: Analyzed are all those included in the mixed model (excludes those with missing covariate data).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | COMPASS | Education Program
Number analyzed (Participants) | 83 | 90
score on a scale
  Baseline | 60.8 (2.2) | 61.2 (2.2)
  12-month follow-up | 74.8 (2.4) | 73.9 (2.6)
Statistical Analysis 1: Comparison: COMPASS vs Education Program; A linear mixed effects model was used to assess the effects of time, group and the interaction of group and time on the outcome. A significant interaction of group and time would indicate that the two groups had significantly different changes in the outcome over time. The model adjusted for race, marital status, living situation, depression, number of days in inpatient rehabilitation, and baseline calendar time; Test type: Superiority; p = 0.76, Mixed Models Analysis — P value shown is for group by time interaction; Mean Difference (Net) = 1.3, 95% CI 2-sided [-7.1 to 9.6] — Between group differences in changes over time (COMPASS vs Education program)

2. Secondary Outcome: Stroke Impact Scale (SIS) - Activities of Daily Living (ADL) Domain
Description: The SIS is a health-related quality of life (HRQoL) measure that quantifies the impact of stroke on a client's life, via questionnaire. The Activities of Daily Living (ADL) domain was used to measure daily activity performance. The scale ranges from 0 to 100, with higher scores indicating less difficulty.
Time Frame: Baseline and 12 months post-stroke
Population: Analyzed are all those included in the mixed model (excludes those with missing covariate data).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | COMPASS | Education Program
Number analyzed (Participants) | 83 | 90
score on a scale
  Baseline | 55.3 (2.3) | 57.0 (2.3)
  12-month follow-up | 66.4 (2.4) | 69.9 (2.6)
Statistical Analysis 1: Comparison: COMPASS vs Education Program; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.60, Mixed Models Analysis — P value shown is for group by time interaction; Mean Difference (Net) = -1.8, 95% CI 2-sided [-8.6 to 5.0] — Between group differences in changes over time (COMPASS vs Education program)

3. Secondary Outcome: In-Home Occupational Performance Evaluation (I-HOPE) - Activity Score
Description: The In-Home Occupational Performance Evaluation (I-HOPE) activity score measures current activity patterns of participants across 44 activities. The score ranges from 0 to 1.0, with a higher score indicating fewer problematic activities for the participant.
Time Frame: Baseline and 12 months post-stroke
Population: Analyzed are all those included in the mixed model (excludes those with missing covariate data).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | COMPASS | Education Program
Number analyzed (Participants) | 82 | 89
score on a scale
  Baseline | 0.73 (0.02) | 0.73 (0.02)
  12-month follow-up | 0.77 (0.02) | 0.78 (0.02)
Statistical Analysis 1: Comparison: COMPASS vs Education Program; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.83, Mixed Models Analysis — P value shown is for group by time interaction; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.06 to 0.05] — Between group differences in changes over time (COMPASS vs Education program)

4. Secondary Outcome: In-Home Occupational Performance Evaluation (I-HOPE) - Performance Score
Description: The In-Home Occupational Performance Evaluation (I-HOPE) performance score is a mean rating of up to 10 participant-prioritized activities on a scale from 1 (unable to perform the activity at all) to 5 (able to perform the activity without difficulty). Higher mean scores indicate better functional ability to perform tasks without difficulty.
Time Frame: Baseline and 12 months post-stroke
Population: Analyzed are all those included in the mixed model (excludes those with missing covariate data).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | COMPASS | Education Program
Number analyzed (Participants) | 78 | 86
score on a scale
  Baseline | 2.42 (0.10) | 2.65 (0.09)
  12-month follow-up | 3.60 (0.10) | 3.44 (0.11)
Statistical Analysis 1: Comparison: COMPASS vs Education Program; A linear mixed effects model was used to assess the effects of time, group and the interaction of group and time on the outcome. A significant interaction of group and time would indicate that the two groups had significantly different changes in the outcome over time. The model adjusted for race, marital status, living situation, depression , number of days in inpatient rehabilitation, and baseline calendar time; Test type: Superiority; p = 0.046, Mixed Models Analysis — P value shown is for group by time interaction; Mean Difference (Net) = 0.39, 95% CI 2-sided [0.01 to 0.77] — Between group differences in changes over time (COMPASS vs Education program)

5. Secondary Outcome: In-Home Occupational Performance Evaluation (I-HOPE) - Satisfaction Score
Description: The In-Home Occupational Performance Evaluation (I-HOPE) satisfaction score is a mean rating of up to 10 participant-prioritized activities on a scale of 1 (not satisfied at all with their performance of the activity) to 5 (very satisfied with their performance of the activity). Higher mean scores indicate more satisfaction with self-rated activity performance.
Time Frame: Baseline and 12-months post-stroke
Population: Analyzed are all those included in the mixed model (excludes those with missing covariate data).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | COMPASS | Education Program
Number analyzed (Participants) | 78 | 86
score on a scale
  Baseline | 2.24 (0.11) | 2.53 (0.11)
  12-month follow-up | 3.56 (0.12) | 3.33 (0.13)
Statistical Analysis 1: Comparison: COMPASS vs Education Program; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.02, Mixed Models Analysis — P value shown is for group by time interaction; Mean Difference (Net) = 0.52, 95% CI 2-sided [0.08 to 0.96] — Between group differences in changes over time (COMPASS vs Education program)

6. Secondary Outcome: In-Home Occupational Performance Evaluation (I-HOPE) - Barrier Severity Score
Description: The In-Home Occupational Performance Evaluation (I-HOPE) barrier severity score is a total sum of barrier ratings (0=independent with/without a device, 1=stand-by assistance needed, 2=minimum assistance needed, 3=moderate assistance needed, 4=maximum assistance needed, 5=no activity ) for all identified barriers across up to 10 prioritized activities. Multiple barriers could be identified for each prioritized activity. Higher sum scores indicate a greater need for assistance/less independence for completion of functional activities. There is no maximum score.
Time Frame: Baseline and 12-months post-stroke
Population: Analyzed are all those included in the mixed model (excludes those with missing covariate data).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | COMPASS | Education Program
Number analyzed (Participants) | 79 | 86
score on a scale
  Baseline | 67.0 (3.6) | 64.4 (3.5)
  12-month follow-up | 30.5 (3.8) | 38.4 (4.1)
Statistical Analysis 1: Comparison: COMPASS vs Education Program; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.07, Mixed Models Analysis — P value shown is for group by time interaction; Mean Difference (Net) = -10.6, 95% CI 2-sided [-21.9 to 0.8] — Between group differences in changes over time (COMPASS vs Education program)

ADVERSE EVENTS:
Time Frame: 1 year post-stroke
Arm/Group | COMPASS | Education Program
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/100
Other Adverse Events (participants affected / at risk) | 0/85 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/20/NCT03485820/Prot_SAP_000.pdf